CLINICAL TRIAL: NCT01671046
Title: Prospective Multicenter Observational Trial to Evaluate Correlation Between Liver Biopsy and Transient Elastography in Liver Fibrosis Assessment and Correlation Between Viral Kinetics and Transient Elastography Evolution During Hepatitis C Treatment in a Population of Chronic HCV Infected Patients
Brief Title: An Observational Study To Assess Liver Fibrosis Stages in Patients With Chronic Hepatitis C Infection
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML27944
Record Dates: First submitted 2012-08-20; First posted 2012-08-23 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Hepatitis C, Chronic
MeSH Terms: conditions — Hepatitis C, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Biopsy of the liver

GROUPS / COHORTS (1):
- Cohort

SUMMARY:
This multi-center, prospective observational study will evaluate the correlation of liver biopsy and transient elastography in liver fibrosis assessment in patients with chronic hepatitis C. Data will be collected for 96 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, >/= 18 years of age
* Chronic Hepatitis C infection (mono-infection or co-infection with human immunodeficiency virus [HIV])
* Detectable level of hepatitis C RNA
* Initiating treatment with pegylated interferon plus ribavirin, or pegylated interferon plus ribavirin, and boceprevir or telaprevir according to local guidelines
* Last liver biopsy performed no later than 3 months prior to enrolment to study

Exclusion Criteria:

* Co-infection with hepatitis B virus
* Previous treatment with pegylated interferon and ribavirin
* Participation in another clinical study in the last 12 months prior to study start

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic hepatitis C
Sampling Method: Probability Sample
Enrollment: 123 (Actual)
Dates: Start 2012-07; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Correlation of liver elasticity with liver biopsy performed no later than 3 months before study start | 24 months
Correlation of liver elasticity evolution with viral kinetics | 24 months

SECONDARY OUTCOMES:
Safety: incidence of adverse events | 24 months
Correlation of liver fibrosis stages with sustained virological response (SVR) | 24 months
Correlation of patients characteristics with sustained virological response | 24 months
Hepatic transient elastography (M-transducer) | 24 months
Hepatic transient elastography (XL-transducer) | 24 months
Correlation of hepatic steatosis score with sustained virological response | 24 months
Correlation of liver steatosis measured by Controlled Attenuation Parameter (CAP) with that obtained by liver biopsy | 24 months
Correlation of liver stiffness of HCV monoinfected patients with HCV/HIV co-infected patients | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (6):
- Brazil (6):
  - Rio de Janeiro, Rio de Janeiro
  - Botucatu, São Paulo
  - Campinas, São Paulo
  - Santo André, São Paulo
  - São Paulo, São Paulo
  - Sorocaba, São Paulo